CLINICAL TRIAL: NCT04778592
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ETX-018810 in Subjects With Lumbosacral Radicular Pain
Brief Title: Efficacy and Safety of ETX-018810 in Subjects With Lumbosacral Radicular Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eliem Therapeutics (UK) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETX-018810-201
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Lumbosacral Radiculopathy

STUDY DESIGN:
Intervention Model Description: Placebo Controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ETX-018810 (Experimental): Drug: ETX-018810 BID for 4 weeks
  Interventions: Drug: ETX-018810
- Placebo (Placebo Comparator): Matching Placebo BID for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETX-018810 — Study Drug
  Arms: ETX-018810
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy and Safety of ETX 018810 in Subjects with Lumbosacral Radicular Pain

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ETX 018810 in Subjects with Lumbosacral Radicular Pain

ELIGIBILITY:
Inclusion Criteria:

* The subject has pain consistent with a diagnosis of chronic lumbosacral radiculopathy due to injury of the lumbosacral nerve root(s)
* The subject reports at least moderate pain intensity at screening.
* The subject's onset of leg pain due to LSRP is at least 3 months
* The subject has a magnetic resonance imaging (MRI) scan that is normal or shows incidental lesions
* The subject has a calculated creatinine clearance ≥30 mL/min
* The subject has clinical laboratory values within normal limits or abnormal values that the investigator deems not clinically significant.
* body mass index (BMI) <40 kg/m2.

Exclusion Criteria:

* The subject has previously undergone back surgery
* The subject is unable to reliably delineate or assess pain by anatomical location/distribution on a body map.
* The subject has a history of peripheral neuropathy, evidence of peripheral neuropathy, or evidence of mononeuropathy in the same limb of LSRP.
* The subject has pain due to infection/abscess, hematoma, or malignancy or other pain that may interfere with the assessment of LSRP in the legs.
* The subject has clinically significant and/or unstable renal, hepatic, hematologic, endocrine, immunologic, inflammatory/rheumatologic, respiratory, or cardiovascular disease that would compromise participation in the study
* The subject has any neurological disease that could interfere with participation in the study (e.g., Huntington's disease, Parkinson's disease, Alzheimer's disease, multiple sclerosis, seizures, epilepsy, stroke).
* The subject has a history or current diagnosis of major psychiatric disorder(s)
* The subject has a has a history of substance abuse or dependence
* The subject has clinically significant abnormal electrocardiogram (ECG) findings
* The subject has received nerve blocks and/or steroid injections for LSRP within the 3 months before screening
* The subject is unwilling or unable to discontinue current medications for LSRP, including topical agents.
* The subject is unable to refrain from using prohibited meds during the study, including: NSAID, antiepileptic drugs, steroids, cannabinoids, or major opioids, antidepressants, muscle relaxants, tramadol, or tapentadol.
* The subject has used prohibited nonpharmacologic therapies, including acupuncture, transcutaneous electrical nerve stimulation, within 30 days the study.
* The subject is currently participating in another or the same clinical study or participated in another clinical study within 3 months before screening
* The subject is pregnant or lactating or not practicing adequate birth control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Delta Clinical Research, Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - DBPS Research LLC, Greenwood Village, Colorado
  - Charter Research, Lady Lake, Florida
  - Cordova Research Institute, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Drug Studies America, Marietta, Georgia
  - Better Health Clinical Research, Newnan, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Anesthesia Research Specialist, Chicago, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Healthcare Research Network, Hazelwood, Missouri
  - Drug Trials America, Hartsdale, New York
  - University of Rochester Translational Pain Research, Rochester, New York
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Meta Medical Research Institute, Dayton, Ohio
  - Clinical Investigations LLC, Edmond, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Precision Spine care, Tyler, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Northwest Clinical Research center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ETX-018810: Drug: ETX-018810 bid
  ETX-018810: Study Drug
- Placebo: Matching Placebo bid
  Placebo: Placebo
Period: Overall Study
Arm/Group | ETX-018810 | Placebo
Started | 75 | 74
Completed | 73 | 70
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: The ITT population included all randomized subjects who received at least one dose of study treatment. One subject randomized to ETX-018810 withdrew consent to participate in the study before receiving their first dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | ETX-018810 | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 61 | 118
  >=65 years | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.29) | 53.8 (10.67) | 54.8 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 36 | 82
  Male | 28 | 38 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 56 | 55 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Daily Pain Score as Derived From the Subject's Responses on the Pain Intensity Numerical Rating Scale (PI-NRS)
Description: Change from baseline in the weekly average of the daily pain score as derived from the subject's responses on the Pain Intensity Numerical Rating Scale (PI-NRS), a 10 point scale from 0 being the least (No Pain) to 10 being the most (Worst Possible Pain).
Time Frame: Baseline to Week 4
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 73 subjects in both the ETX-018810 and Placebo groups. All subjects in this population were included in the statistical analysis comparing the groups. However, the descriptive statistics for Week 4 only include those subjects who had measurements at Baseline and Week 4 (72 and 70 subjects, respectively).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 72 | 70
units on a scale | -1.49 (1.735) | -1.65 (1.760)
Statistical Analysis 1: Comparison: ETX-018810 vs Placebo; Test type: Superiority; p = 0.4549, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.36 to 0.79], Standard Error of Mean 0.291

2. Secondary Outcome: Number of Subjects With ≥50% Reduction From Baseline to Weeks 1, 2, 3,and 4 in the Weekly Average of the Daily Pain Score
Description: Change in the weekly average of the daily pain score as derived from the subject's responses on the Pain Intensity Numerical Rating Scale (PI-NRS), a 10 point scale from 0 being the least (No Pain) to 10 being the most (Worst Possible Pain).
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 73 subjects in both the ETX-018810 and Placebo groups. Not all subjects had assessments at each week.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Week 1: number analyzed (Participants) | 72 | 73
  Week 1 | 4 | 3
  Week 2: number analyzed (Participants) | 73 | 71
  Week 2 | 9 | 8
  Week 3: number analyzed (Participants) | 73 | 72
  Week 3 | 12 | 17
  Week 4: number analyzed (Participants) | 72 | 70
  Week 4 | 14 | 17

3. Secondary Outcome: Number of Subjects With a ≥30% Reduction From Baseline to Weeks 1, 2, 3, and 4 in the Weekly Average of the Daily Pain Score
Description: as for outcome 2
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Week 1: number analyzed (Participants) | 72 | 73
  Week 1 | 9 | 17
  Week 2: number analyzed (Participants) | 73 | 71
  Week 2 | 18 | 19
  Week 3: number analyzed (Participants) | 73 | 72
  Week 3 | 22 | 28
  Week 4: number analyzed (Participants) | 72 | 70
  Week 4 | 28 | 29

4. Secondary Outcome: Change in the Weekly Average of the Daily Pain Score From Baseline to Weeks 1, 2, and 3
Description: as for outcome 2
Time Frame: Baseline to Weeks 1, 2, and 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 73
score on a scale
  Week 1: number analyzed (Participants) | 72 | 73
  Week 1 | -0.66 (1.079) | -0.85 (0.994)
  Week 2: number analyzed (Participants) | 73 | 71
  Week 2 | -1.04 (1.479) | -1.15 (1.429)
  Week 3: number analyzed (Participants) | 73 | 72
  Week 3 | -1.28 (1.575) | -1.49 (1.606)

5. Secondary Outcome: Change From Baseline to Week 4 for Worst Pain
Description: The Brief Pain Inventory (BPI) includes a 'worst pain' severity scale. Subjects rate their worst pain in the last 24 hours on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline and Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 74 subjects in both the ETX-018810 and Placebo groups. Not all subjects had a BPI assessment at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 72
score on a scale | -1.73 (2.206) | -1.74 (1.861)

6. Secondary Outcome: Number of Subjects With a PGI-C Response (Defined as "Much Improved" or "Very Much Improved") at Week 4
Description: The Patient Global Impression - Change (PGI-C) is the patient-reported counterpoint to the CGI-C (Guy, 1976). The qualitative assessment of meaningful change is determined by the patient in response to the question, "Compared to your condition at the beginning of treatment, how much has your condition changed?" Scores are as follows: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse.
Time Frame: Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 74 subjects in both the ETX-018810 and Placebo groups. Not all subjects had a PGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 74 | 73
Participants | 23 | 25

7. Secondary Outcome: Number of Subjects With a CGI-C Response (Defined as "Much Improved" or "Very Much Improved") at Week 4
Description: The Clinical Global Impression - Change (CGI-C) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to the baseline state at the beginning of the intervention. The rater selects one response based on the following question, "Compared to your patient's condition at the beginning of treatment, how much has your patient changed?" Scores are as follows: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse.
Time Frame: Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 74 subjects in both the ETX-018810 and Placebo groups. Not all subjects had a CGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 74 | 73
Participants | 21 | 24

8. Secondary Outcome: Change in the Weekly Average of the Daily Sleep Score on the DSIS From Baseline to Weeks 1, 2, 3, and 4
Description: The Daily Sleep Interference Scale (DSIS) is an 11-point response scale that quantifies sleep interference due to pain. It is a single-item measure that is completed once daily, upon awakening, to accurately capture variability in sleep interference due to pain on a daily basis, thus minimizing recall bias. Patients are asked to select the number that best described how much their pain has interfered with their sleep during the last 24 hours on a scale from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep).
  The subjects were to record the value that most closely corresponded to their sleep interference over the last 24 hours in the eDiary once daily, in the morning (when the first dose of investigational medication is taken), during the baseline and 4-week treatment periods.
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 73
score on a scale
  Week 1: number analyzed (Participants) | 72 | 73
  Week 1 | -0.87 (1.279) | -0.81 (1.114)
  Week 2: number analyzed (Participants) | 73 | 71
  Week 2 | -1.14 (1.576) | -1.18 (1.366)
  Week 3: number analyzed (Participants) | 72 | 71
  Week 3 | -1.41 (1.697) | -1.51 (1.520)
  Week 4: number analyzed (Participants) | 72 | 71
  Week 4 | -1.59 (1.676) | -1.53 (1.706)

9. Secondary Outcome: Change in BPI - Interference Scale From Baseline to Week 4
Description: The Brief Pain Inventory (BPI) interference score measures how much pain has interfered with seven daily activities scored on a scale from 0 (does not interfere) to 10 (completely interferes). It is scored as the mean of the seven interference items.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 72
score on a scale | -1.68 (1.967) | -1.94 (1.954)

10. Secondary Outcome: Change in the BPI - Pain Scale From Baseline to Week 4
Description: The Brief Pain Inventory (BPI) pain score is a composite of 4 items assessing pain severity (worst, least, average and right now). Subjects rate their pain in the last 24 hours on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). It is scored as the mean of the four pain items.
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 72
score on a scale | -1.70 (1.974) | -1.57 (1.588)

11. Secondary Outcome: Change in the RMDQ From Baseline to Week 4
Description: The modified Roland-Morris Disability Questionnaire (RMDQ) is a self-administered, 24-question physical disability measurement assessment that evaluates the effect of back pain on functioning. Each question requires a "yes" or "no" answer; 1 point is scored for each positive response. The total scores are determined on a scale of 0 ("no disability") to 24 ("severe disability").
Time Frame: Baseline to Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 74 subjects in both the ETX-018810 and Placebo groups. Not all subjects had a RMDQ assessment at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 73 | 71
score on a scale | -2.10 (3.637) | -2.31 (4.367)

12. Secondary Outcome: Change in the Daily Amount of Acetaminophen Use From Baseline to Week 4
Description: The daily amount of acetaminophen (rescue medication) used (mg per day).
Time Frame: Treatment period: 4 weeks
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 73 subjects in both the ETX-018810 and Placebo groups. Three subjects were excluded due to implausible records in the subject's diary.
Measure: Median (Inter-Quartile Range); unit: mg per day
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 72 | 71
mg per day | 0 [-99.4 to 0] | 0 [-177.3 to 9.3]

ADVERSE EVENTS:
Time Frame: 9 weeks (up to 4 week screening period, 4 week treatment period, & 1 week follow up period)
Arm/Group | ETX-018810 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/74
Other Adverse Events (participants affected / at risk) | 11/74 | 15/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETX-018810 (N=74) | Placebo (N=74)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETX-018810 (N=74) | Placebo (N=74)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the PI will provide the sponsor with a copy of any proposed communication at least 90 days in advance of the proposed submission or presentation date. Within this 90 day period, the sponsor will review the communication to determine whether it contains any sponsor Confidential Information, or whether the sponsor desires to file patent applications on subject matter contained therein, and to ensure the accuracy of the information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT04778592/Prot_SAP_000.pdf